CLINICAL TRIAL: NCT03878654
Title: Trial of Tauroursodeoxycholic Acid (TUDCA) in Asthma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: IRB protocol violations
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, David Kaminsky, MD, Professor of Medicine, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UVermont
Record Dates: First submitted 2019-01-21; First posted 2019-03-18 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — ursodoxicoltaurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tauroursodeoxycholic Acid (Experimental): TUDCA 1750 mg daily for 12 weeks
  Interventions: Drug: Tauroursodeoxycholic Acid

INTERVENTIONS:
Drug: Tauroursodeoxycholic Acid — Naturally occurirng bile acid
  Other Names: Taurolite

SUMMARY:
Asthma is a chronic lung disease that affects millions of people worldwide, including both children and adults. The cause of asthma is not known, but asthma is strongly associated with inflammation of the airways, often caused by allergies. In order to control this inflammation, most people with asthma are treated with inhaled medications that contain steroids. These medications do a good job of helping most people with asthma feel better. However, these medications are expensive, have side effects, and do not control symptoms in all people with asthma. Recently basic science research colleagues have shown that inflammation due to allergies can be reduced in experimental animals by a naturally occurring bile acid. Bile acids are chemicals made in the liver that are involved in maintaining healthy digestion of fat. Since bile acids are made by our bodies, they have become popular as over the counter supplements that are thought to be important in promoting a healthy liver and metabolism. Interestingly, other research has shown that bile acids may help patients with neurological disease and diabetes.

Given all of this information, the investigators propose that a specific bile acid called tauroursodeoxycholic acid (TUDCA) may be helpful in patients with asthma. Before studying this in a clinical trial, the current study is designed to demonstrate that people with asthma can take TUDCA safely and that it doesn't hurt their asthma. The study will involve inviting 12 patients with mild asthma to take TUDCA daily for 12 weeks. During this time the investigators will closely monitor them for any side effects and check their blood and breathing capacity for any signs of detrimental effects. In addition, the investigators will collect cells that line the nose, which are thought to be similar to cells in the airways of the lungs, to see if TUDCA is having any beneficial effects on inflammation. In order to ensure the use of high quality TUDCA, which may or may not be true of over the counter supplements, the investigators have asked the company that is supplying TUDCA for the studies mentioned previously involving neurological disease and diabetes to supply the drug; the brand name is Taurolite. In addition, even though TUDCA is available over the counter, in order to use it for research, the FDA has to approve this use. Accordingly, the investigators have applied for and received permission (IND) from the FDA to use Taurolite for this study.

DETAILED DESCRIPTION:
Study Design: This study will be a Phase 1, pre-post intervention trial in patients with asthma who will be treated with TUDCA 1750 mg per day for 12 weeks. The investigators have obtained TUDCA from Bruschettini (http://www.bruschettini.com), which is an authorized Italian pharmaceutical company that can provide validation of the drug's manufacture and purity. Bruschettini markets TUDCA under the brand name Taurolite. The investigators have received an IND from the FDA for use of Taurolite in this study (see document).

Protocol: All participants will undergo an initial screening visit by telephone to determine. Participants will then present to the Vermont Lung Center in Colchester for 2 study visits, during which the following testing and information will be obtained:

Visit 1 (Baseline)

* Demographics: age, sex, height, weight
* Concomitant medical problems and medications
* Asthma control by ACT
* Lung function testing: spirometry (FEV1, FVC, FEV1/FVC) (43), forced oscillation technique (FOT) (R5, R20, X5, AX, Fres) (44)
* Fraction of exhaled nitric oxide (FeNO) as a general measure of eosinophilic inflammation(45)
* Blood sample collection for routine chemistries (10 cc), and for analysis of serum markers of inflammation (10 cc).
* Nasal brushing for collection of epithelial cells for analysis of serum markers of ER stress and UPR The participant will then receive a supply of medication, TUDCA 250 mg, to be taken 500 mg with breakfast, 500 mg with lunch, 750 mg with dinner, daily, for 12 weeks.

The participant will also receive a daily diary to use to record daily symptoms of asthma and any side effects, as well as compliance with taking the medication.

Visit 2 (Week 4) and Visit 3 (Week 8)

* Review of diary for side effects, adverse events
* Asthma control by ACT, spirometry, FeNO
* Blood for routine chemistries as part of ongoing safety monitoring Visit 4 (Week 12) All testing as listed for Visit 1 will be repeated, with collection of any remaining drug and all diary data.

Telephone Calls (Weeks 2,6,10) The investigators will call participants every 2 weeks in between study visits to assess tolerability and remind participants to complete their daily diaries. The investigators will use a standardized questionnaire for study coordinators to use during each assessment by telephone to determine whether there have been any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 and older, with a physician diagnosis of asthma
* Current non-smoker with < 10 pack-years smoking history and no smoking within the last year
* Stable asthma control over the last 3 months as defined by Asthma Control Test (ACT) ≥ 20 (40)
* Stable asthma medication regimen over the last 3 months
* FEV1 ≥ 70% predicted

Exclusion Criteria:

* Current smoking or ≥10 pack-years of smoking or any smoking within the last year
* Poor asthma control as defined by ACT< 20
* Exacerbation of disease within previous 4 weeks
* Recent upper respiratory infection within last 4 weeks
* Acute or chronic rhinosinusitis
* Use of chronic nasal corticosteroids, or any use of nasal corticosteroids during the study
* Concomitant heart, lung or GI disease (liver, peptic ulcer) that would potentially jeopardize the safety of the participant or interfere with interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
AST | 12 weeks
  Liver toxicity by AST
ALT | 12 weeks
  Liver toxicity by ALT
alkaline phosphatase | 12 weeks
  Liver toxicity by alkaline phosphatase
total bilirubin | 12 weeks
  Liver toxicity by total bilirubin
BUN | 12 weeks
  Renal toxicity by BUN
creatinine | 12 weeks
  renal function by creatinine
CBC | 12 weeks
  Hematology toxicity by CBC
total cholesterol | 12 weeks
  Lipid toxicity by total cholesterol
LDL | 12 weeks
  Lipid toxicity by LDL
HDL | 12 weeks
  Lipid toxicity by HDL
triglycerides | 12 weeks
  Lipid toxicity by triglycerides
symptom diary | 12 weeks
  symptoms and side effects

SECONDARY OUTCOMES:
ACT score | 12 weeks
  Asthma control by ACT score
spirometry | 12 weeks
  Lung function by spirometry
forced oscillation | 12 weeks
  Lung function by spirometry
FeNO | 12 weeks
  Airway eosinophilic inflammation by FeNO
peripheral eosinophil count | 12 weeks
  Allergic inflammation by peripheral eosinophil count
IgE | 12 weeks
  Allergic inflammation by peripheral eosinophil count
HSPA5 (GRP78) | 12 weeks
  Markers of ER stress in nasal epithelium - HSPA5 (GRP78)
DDIT (CHOP) | 12 weeks
  Markers of ER stress in nasal epithelium - DDIT (CHOP)
PDIA3 | 12 weeks
  Markers of ER stress in nasal epithelium - PDIA3
XBP1 | 12 weeks
  Markers of ER stress in nasal epithelium - XBP1
serum periostin | 12 weeks
  Allergic inflammation by serum periostin
CCL-20 | 12 weeks
  Allergic inflammation by CCL-20
IL-4 | 12 weeks
  Allergic inflammation by IL-4
IL-5 | 12 weeks
  Allergic inflammation by IL-5
IL-13 | 12 weeks
  Allergic inflammation by IL-13
IL-17A | 12 weeks
  Allergic inflammation by IL-17A

CONTACTS AND LOCATIONS:
Overall Officials: David Kaminsky, MD, Principal Investigator — University of Vermont
Locations (1):
- Vermont Lung Center, Colchester, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siddesha JM, Nakada EM, Mihavics BR, Hoffman SM, Rattu GK, Chamberlain N, Cahoon JM, Lahue KG, Daphtary N, Aliyeva M, Chapman DG, Desai DH, Poynter ME, Anathy V. Effect of a chemical chaperone, tauroursodeoxycholic acid, on HDM-induced allergic airway disease. Am J Physiol Lung Cell Mol Physiol. 2016 Jun 1;310(11):L1243-59. doi: 10.1152/ajplung.00396.2015. Epub 2016 May 6. PMID 27154200